CLINICAL TRIAL: NCT06410326
Title: Mapping the Longitudinal, Multidimensional Impact of MS in Relation to Variables Indicative of Neurological Reserve
Acronym: Resilience
Status: Completed | Type: Observational
Sponsor: National MS Center Melsbroek (Other)
Collaborators: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Marie D'hooghe, Prof Dr D'hooghe, National MS Center Melsbroek
Other Study IDs: Resilience
Record Dates: First submitted 2024-04-04; First posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Some MS patients quickly accumulate neurological deficits, while others remain well for decades. Even though associations with age, sex, health behaviors, comorbidities and social determinants of health are widely acknowledged, the clinical heterogeneity in MS is poorly understood and variables with a robust prognostic value are lacking. Recent data suggest a key role for resilience in the central nervous system, potentially supporting the concept of neurological reserve in MS.

DETAILED DESCRIPTION:
The first phase of the study will take place at the National MS Center Melsbroek (NMSC). All data from the EDMUS database, a single center database at the NMSC, will be exported and checked (quantity, quality) aiming to come to a well-organized MS data structure. This MS register will be completed with volume data (intracranial, spinal canal) in a subset of patients. As a substantial number of MS patients are followed over the long-term in the MS center, the investigators expect to have longitudinal data well beyond a disease duration of 10 years at least for part of the patients. Following the export and cleaning phase of the data, the investigators will come to the basic descriptive statistics. This allows us to have an overview of all data and determine the most appropriate baseline variables or covariates as well as to define the most appropriate outcome variables. Multivariable regression analysis will be used to predict the value of outcome variables based on the independent variables whose values are known. In view of the relevance of age and disease duration in the context of MS disability and progression, time-to-event analysis will be performed, with the time to reach irreversible milestones of ambulatory disability as outcome.

In case of associations, the second phase of the study will be initiated for further analysis at the AIMS research group, VUB. At the AIMS group, VUB, the potential of false positive findings will be addressed using more sophisticated approaches (splitting cohorts in exploratory and discovery cohort, or cross-fold validation).

ELIGIBILITY:
Inclusion Criteria:

diagnosis of MS needs to be based on diagnostic criteria valid at the time of data entry and confirmed during follow up

Exclusion Criteria:

* Neuromyelitis Optica diagnosis, AQ4 positive or MOG positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple Sclerosis patients followed in the National MS center Belgium
Sampling Method: Non-Probability Sample
Enrollment: 2600 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
EDSS | 2 years
  The EDSS ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability. In the lower part of its range, the EDSS score predominantly reflects the result of the examination by a neurologist, primarily a measure of impairment in eight functional systems (FS). In the middle part of its range, the EDSS score is primarily a measure of ambulation ability. At the higher end, upper limb and bulbar function as well as the ability to accomplish activities of daily living determine the score. The EDSS is considered to be an ordinal scale. The point estimates of the central tendency should be presented as median values and the measures of dispersion as interquartile ranges (Uitdehaag B, 2014).
  According to Havardova et al, MSJ 2017, the following disease severity groups can be distinguished:
  Mild EDSS 0-3 Moderate EDSS 4-6.5 Severe EDSS 7-9
Functional tests | 2 years
  Functional tests of upper limbs (9-HPT) and lower limbs (25FWT) are measured in seconds. Higher scores indicate a worse function. A 20% change of the scores is considered to be a reasonable cutoff value for reliably detecting a clinically meaningful change.
Cognitive tests | 2 years
  Cognitive screening tests include the PASAT (till 2015) and the SDMT (since 2015). The results are corresponding to the number of correct answers in a fixed time frame. Higher scores indicate a better function. The tests were usually performed on a yearly basis to limit learning effects.
The EQ-Visual Analog Score (EQ-VAS) | 2 years
  The EQ-Visual Analog Score (EQ-VAS) records the patient's self-rated health on a vertical visual analogue scale, a kind of 'thermometer' where the endpoints are labelled 'The best health you can image' (endpoint 100 at the top) and 'The worst health you can image' (endpoint 0 at the bottom). The patient is asked to draw a line from the box marked 'Your health status today' to the appropriate point on the 'thermometer' scale. The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement.
  The 5-level EQ-5D version (EQ-5D-5L) was introduced by the EuroQol Group in 2009 to improve the instrument's sensitivity and to reduce ceiling effects, as compared to the EQ-5D-3L. Five questions assessing five domains (mobility, self-care, usual activity, pain/discomfort, anxiety/depression) are included. A single index value can be generated.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationaal Multiple Sclerose Centrum Melsbroek, Melsbroek, Vlaams-Brabant, Belgium